CLINICAL TRIAL: NCT04808310
Title: QUantitative Flow Ratio Or Angiography for the assessMent of nOn-culprit Lesions
Acronym: QUOMODO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Tommaso Gori, Clinical Professor, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-15296
Record Dates: First submitted 2021-03-17; First posted 2021-03-22 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to one of the two study arms. Randomization will be done by using a computer-generated random sequence (Medcalc, Mariakerke, BE).
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and outcome assessors will be blinded to the randomization group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angiography (Active Comparator): The indication to further coronary intervention will be based on angiographic diameter stenosis.
  Interventions: Diagnostic Test: Assessment of angiographic severity of the stenosis
- Quantitative flow ratio (QFR) (Experimental): The indication to further coronary intervention will be based on QFR.
  Interventions: Device: Quantitative flow ratio

INTERVENTIONS:
Device: Quantitative flow ratio — Quantitative flow ratio (QFR) is a computer method that estimates the hemodynamic relevance of a coronary stenosis based on three-dimensional quantitative coronary angiography (3D QCA)
  Arms: Quantitative flow ratio (QFR)
Diagnostic Test: Assessment of angiographic severity of the stenosis — The indication to coronary stent intervention will be based on angiography
  Arms: Angiography

SUMMARY:
The aim of this study is to study whether the use of complex 3-dimensional assessment of the severity of a stenosis improves angina and in general cardiovascular outcomes in patients who have residual intermediate coronary artery stenosis following an acute coronary syndrome (ACS) treated with percutaneous coronary intervention (PCI).

Goals of the study are:

* To investigate whether decision-making based on quantitative flow reserve (QFR) is associated with a decrease in angina 3 months after an ACS
* To investigate whether use of QFR is associated with an improved prognosis.

DETAILED DESCRIPTION:
The study is a single-center, randomized superiority trial to compare two strategies for the assessment of the hemodynamic relevance of coronary lesions.

The primary analysis will be on the per-protocol principle (i.e. including all patients who are not protocol violators). A separate analysis will be performed on an intention-to-treat basis (i.e. all randomized patients randomized to a treatment arm).

Primary endpoint 1. Angina questionnaire

Secondary endpoints:

Number and % of patients undergoing PCI

Seattle Angina Questionnaire

* SAQ Physical limitation scale
* SAQ angina stability scale
* SAQ angina frequency scale
* SAQ quality of life
* SAQ Treatment Satisfaction Disease perception scale Follow-up (3 and 12 months) - Patient-oriented composite endpoint (death, myocardial infarction, unplanned revascularization) and its components.

ELIGIBILITY:
Inclusion Criteria:

* Successfully treated acute coronary syndrome
* At least one additional intermediate stenosis (>30% and <90%).
* Patient ≥18 years old

Exclusion Criteria:

* Stenoses or patients a priori not amenable to treatment with PCI (at the discretion of two interventional cardiologists - e.g. patients with limited life expectancy, stenosis in very small vessels, very diffuse disease with complex/very calcified stenosis requiring surgery etc).
* Persistent symptoms or evidence of ischemia requiring intervention of the non-culprit lesion.
* Any contraindication to PCI according to guidelines
* An ACS in the period following the index ACS and randomization
* TIMI (Thrombolysis in Myocardial Infarction) flow grade < 3 in the culprit vessel
* Presence of thrombus in the non-culprit lesion
* Participation in another randomized interventional study interfering with the present protocol
* Patient unable to give informed consent
* Women of child-bearing potential or lactating
* Previous coronary artery bypass surgery CABG
* Recent (within 30 days) unsuccessful PCI
* Decompensated congestive heart failure (CHF) or hospitalization due to CHF during the last 3 months
* Left ventricular ejection fraction <30%
* Severe chronic obstructive pulmonary disease (COPD)
* Severe valvular heart disease
* FFR (or RFR, iFR etc) assessment of non-culprit lesions at the time of the index procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
Patient-oriented combined endpoint (clinical endpoint) | 12 months
  composite of patient-oriented events and significant angina (all-cause death, non fatal myocardial infarction including type 1, 2, 4, unplanned hospitalization for angina or heart failure, unplanned revascularization, SAQ<90)
Functional endpoint | Upon randomization and following QFR assessment
  Proportion of patients assigned to medical treatment in the two groups (QFR vs. Reference)

SECONDARY OUTCOMES:
Seattle angina questionaire summary score | 12 months
  Angina severity as assessed by the Seattle Angina Questionnaire (SAQ, score of 0 to 100, where higher scores indicate better function (eg, less physical limitation, less angina, and better quality of life))
Seattle angina questionaire summary score | 3 months
  Angina severity as assessed by the Seattle Angina Questionnaire (SAQ, score of 0 to 100, where higher scores indicate better function (eg, less physical limitation, less angina, and better quality of life))
Unplanned admission | 12 months
  Incidence of unplanned hospital admission for angina
Patient-oriented composite endpoint | 3 months
  Patient-oriented composite endpoint (death, myocardial infarction, unplanned revascularization).
Patient-oriented composite endpoint | 12 months
  Patient-oriented composite endpoint (death, myocardial infarction, unplanned revascularization).

CONTACTS AND LOCATIONS:
Locations (1):
- Center of Cardiology, Cardiology I, university hospital Mainz, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ullrich-Daub H, Olschewski M, Schnorbus B, Belhadj KA, Kohler T, Vosseler M, Munzel T, Gori T. Quantitative flow ratio or angiography for the assessment of non-culprit lesions in acute coronary syndromes, a randomized trial. Clin Res Cardiol. 2025 Jun;114(6):729-737. doi: 10.1007/s00392-024-02484-5. Epub 2024 Jul 9. PMID 38980329
- [Derived] Ullrich H, Olschewski M, Belhadj KA, Munzel T, Gori T. Quantitative Flow Ratio or Angiography for the Assessment of Non-culprit Lesions in Acute Coronary Syndromes: Protocol of the Randomized Trial QUOMODO. Front Cardiovasc Med. 2022 Apr 4;9:815434. doi: 10.3389/fcvm.2022.815434. eCollection 2022. PMID 35445090